CLINICAL TRIAL: NCT00123760
Title: A Phase I/II, Phase III and Extended Phase III Study of 18F-Fluorodeoxyglucose (FluGlucoScan) in Patients With Cancer or Suspected Cancer
Brief Title: Study of 18F-Fluorodeoxyglucose (FluGlucoScan) in Patients With Cancer or Suspected Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SP-11-0035/DX-FDG-001/21221
Record Dates: First submitted 2005-07-22; First posted 2005-07-26 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2012-03

CONDITIONS: Brain Neoplasms; Lung Neoplasms; Thyroid Neoplasms; Colorectal Neoplasms; Lymphoma
Keywords: Positron-Emission Tomography; Fluorodeoxyglucose F18; Tomography scanners, X-Ray computed
MeSH Terms: conditions — Brain Neoplasms; Lung Neoplasms; Thyroid Neoplasms; Colorectal Neoplasms; Lymphoma | interventions — Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Positron Emission Tomography (PET) scan

SUMMARY:
Positron Emission Tomography (PET) is a specialised nuclear medicine procedure that uses positron emitting radiolabeled tracer molecules to measure biological activity. The most common of these radiolabeled tracers is 18F-fluorodeoxyglucose (18F-FDG), which is used to determine abnormal glucose metabolism in tumours and other sites. It has general applications in all areas where abnormal glucose metabolism may be present including in circumstances such as differentiating the tumour from scar tissue; evaluating the presence of the tumour in light of rising tumour markers and normal morphological imaging techniques; and assessing response to therapy where other techniques are deemed to be unhelpful. The Cross Cancer Institute (CCI) has recently been funded to establish a PET centre, and this study will prove the effectiveness of PET scanning in the Canadian health care environment and validate the data that have been developed in other jurisdictions in specific oncologic indications.

DETAILED DESCRIPTION:
Background

Positron Emission Tomography (PET) is a specialised Nuclear Medicine procedure that uses positron emitting radiolabeled tracer molecules to measure biological activity. The commonest of these radiolabeled tracers is 18F-Fluorodeoxyglucose (18F-FDG), which is used to determine abnormal glucose metabolism in tumours and other sites. It has general applications in all areas where abnormal glucose metabolism may be present including circumstances such as differentiating tumour from scar tissue, evaluating the presence of tumour in the light of rising tumour markers and normal morphological imaging techniques and assessing response to therapy where other techniques are deemed to be unhelpful.

The Cross Cancer Institute has recently been funded to establish a PET centre that will establish a research programme to prove the effectiveness of PET scanning in the Canadian health care environment and validate the data that have been developed in other jurisdictions in specific oncologic indications.

Objectives

Primary Objectives - The objectives of the clinical trial are to (a) demonstrate the safety of 18F-FDG synthesised from cyclotron produced radiofluoride in the Coincidence Technologies automated synthesis unit (ASU) in the Edmonton PET Centre facility and (b) confirm the diagnostic effectiveness of 18F-FDG in subjects with known or suspected oncologic disease and to compare this with values published in the literature.

Secondary Objectives - The secondary objectives of the clinical trial are to confirm the general utility and value of 18F-FDG imaging of abnormal glucose metabolism in oncologic applications, particularly with respect to Canadian practice.

Study Design

The proposed clinical trial will be a combined Phase I/II, Phase III, extended Phase III (Phase I/II,III,exIII), diagnostic imaging, controlled, open label, single site, clinical trial in a broad cross-section of CCI patients, including patients with Hodgkin and non-Hodgkin lymphoma, colorectal cancer, breast cancer, melanoma, head and neck cancers, PRUNK, esophageal cancer, thyroid cancer, NSCLC, SCLC, neuroendocrine tumours, and patients with CNS tumours where conventional imaging methods have failed to yield a diagnostic answer.

Each patient will usually receive a single IV injection of 18F-FDG. Imaging will be conducted 30 to 60 minutes after an average injection of 200 - 300 MBq of 18F-FDG in hydrated, fasted patients. Images will be collected for 40 to 60 minutes in 5 - 7 body positions (total counts 5 to 15 million). For the Phase I/II study, images will be interpreted by a single experienced Nuclear Medicine physician with regard to normal physiological uptake of 18F-FDG. For the Phase III study, images will be interpreted independently by two experienced Nuclear Medicine physicians with regard to normal physiological uptake of 18F-FDG. The location and intensity of abnormal 18F-FDG uptake will be noted and correlated with clinical findings, surgical or biopsy results or with conventional imaging techniques, as available. The image review will be supplemented with access to clinical and conventional imaging data in the Phase I/II study. In the Phase III study all images will be reviewed independently by one physician blinded to all clinical data except the primary diagnosis and by one physician with access to all relevant clinical information. In the extended Phase III protocol the images will be interpreted by a single physician with access to relevant clinical information

Statistical Analyses

Sample Size

The Phase I/II stage will enroll 20 subjects without regard for tumour type. The Phase III stage will enroll approximately 300 subjects and the extended Phase III stage will enroll approximately 3000 subjects with the approximate distribution by tumour type as follows:

Tumour Type Phase III:Extended Phase III

* Brain 10:100
* Colorectal 33:330
* Breast 21:210
* Lung (NSCLC & SCLC) 130:1300
* Lymphoma (Hodgkin's and non-Hodgkin's) 22:220
* Head & Neck 16:160
* Neuroendocrine 10:100
* Thyroid 29:290
* Melanoma 15:150
* PRUNK 14:140

Within each cancer subgroup in the Phase III stage, where disease status confirmation is available, the sensitivity (true positive outcomes/true positive outcomes + false negative outcomes) and positive predictive value (true positive outcomes/true positive outcomes + false positive outcomes) will be calculated on a per patient basis. The general criteria for assessment of comparability is that the study group sensitivity percent and positive predictive value percent values have a difference of not less than 15 percent from the appropriately matched literature values. For subgroups with significant patient numbers statistical analysis of comparability will be undertaken.

Criteria for Evaluability of Study Subject Data All subjects enrolled in the Phase I/II stage of the trial will be evaluated for safety. All subjects enrolled in the Phase III and extended Phase III study will be evaluated for safety and efficacy.

Study Population

Number of Subjects to be Studied Phase I/II stage: ~ 20 Phase III stage: ~ 300 Extended Phase III stage: ~ 3000 Some variation in the patient numbers studied is anticipated in the Phase III and extended Phase III depending on local conditions and timing.

Inclusion Criteria for Selection of Study Subjects

Patients will be included in the study if they meet all of the following general criteria.

1. Male or female.
2. Known or suspected primary or metastatic tumours.
3. Age greater than or equal to 15
4. If female of child-bearing potential, a reliable method of contraception must be combined with a negative pregnancy test before entering the study (contraception must be used for 1 month after the last administration of 18F-FDG). If male, a barrier method of contraception should be used for up to 1 month after the last administration of 18F-FDG.
5. Able and willing to follow instructions and comply with the protocol.
6. Provide written informed consent prior to participation in the study.
7. Karnofsky Performance Scale Score 60-100.

Exclusion Criteria

Patients will be excluded from the study if they meet any of the following criteria:

1. significant renal impairment (serum creatinine > 200 µmol/L).
2. Coagulopathy (prothrombin time [PT] or activated partial thromboplastin time [APTT] >1.5 times control).
3. Significant Thrombocytopenia (platelet count < 75,000/mm3).
4. Granulocytopenia (absolute neutrophil count < 1,000/mm3).
5. Blood glucose level Significant liver function impairment (total bilirubin > 2.0 mg/dL; AST or ALT > 3 times the upper limit of normal) or greater than 10.
6. Presence of a severe infection.
7. Having had surgery or radiotherapy within 10 days of the planned imaging study.
8. Nursing or pregnant females.
9. Age less than 15.

ELIGIBILITY:
Inclusion Criteria:

* Male or female. (If female of child-bearing potential and outside of the window of 10 days since the last menstrual period, a negative serum or urine pregnancy test is required.)
* Known or suspected primary or metastatic tumours
* Age equal to or greater than 15 years
* Able and willing to follow instructions and comply with the protocol
* Provide written informed consent prior to participation in this study
* Karnofsky Performance Scale score 60-100

Exclusion Criteria:

* Nursing or pregnant females
* Presence of a severe infection
* Age less than 15 years
* Having had surgery or radiotherapy within 10 days of the planned imaging study

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10838 (Actual)
Dates: Start 2004-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To demonstrate the safety of 18F-FDG synthesized from cyclotron produced radiofluoride in the Coincidence Technologies automated synthesis unit (ASU) in the Edmonton PET Centre facility | One Year

SECONDARY OUTCOMES:
To confirm the diagnostic effectiveness of 18F-FDG in subjects with known or suspected oncologic disease and compare this to literature values | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Alexander McEwan, MB, MSc, MD, FRCP, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada